CLINICAL TRIAL: NCT02642380
Title: Different Cycles of High-dose Dexamethasone for Initial Management of Primary Immune Thrombocytopenia (ITP): a Prospective, Randomized Controlled Trial
Brief Title: Different Cycles of High-dose Dexamethasone for Initial Management of Primary Immune Thrombocytopenia (ITP)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Principal Investigator, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: High-dose dexamethasone
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2015-12

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; high-dose dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4 cycles (Experimental): Oral administration of dexamethasone 40 mg for four consecutive days every 14 days for 4 courses
  Interventions: Drug: Dexamethasone (4 cycles)
- 1 cycle (Active Comparator): Oral administration of dexamethasone 40 mg for four consecutive days
  Interventions: Drug: Dexamethasone (1 cycle)

INTERVENTIONS:
Drug: Dexamethasone (4 cycles) — dexamethasone 40mg daily for 4 consecutive days every 14 days for 4 courses
  Other Names: DXM 4
  Arms: 4 cycles
Drug: Dexamethasone (1 cycle) — dexamethasone 40mg daily for 4 consecutive days
  Other Names: DXM 1
  Arms: 1 cycle

SUMMARY:
The project was organized by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of different cycles of high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, randomized, controlled trial of 200 primary ITP adult patients from 11 medical centers in China. One part of the participants are randomly selected to receive four cycles of high-dose dexamethasone (given orally at a dose of 40mg per day for 4 consecutive days every 14 days for 4 cycles), comparing the others with one cycle (given orally at a dose of 40 mg per day for 4 consecutive days).

Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of different cycles of high-dose dexamethasone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count <30 * 10^9/L, and with bleeding manifestations.
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
sustained response to treatment | 6 months after treatment started
  percentage of patients maintaining PLT count over 30*10^9 without bleeding

SECONDARY OUTCOMES:
Evaluation of early response | 2 months after treatment started
  Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD, PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China